CLINICAL TRIAL: NCT04125927
Title: Open-label, Single-arm, Multicenter Study to Assess the Safety of Cystadrops® in Pediatric Cystinosis Patients From 6 Months to Less Than 2 Years Old
Brief Title: Cystadrops in Pediatric Cystinosis Patients From Six Months to Less Than Two Years Old (SCOB2)
Acronym: SCOB2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYT-C2-001
Record Dates: First submitted 2019-10-03; First posted 2019-10-14 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Cystinosis
MeSH Terms: conditions — Cystinosis | interventions — Cysteamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-label arm (Experimental)
  Interventions: Drug: Mercaptamine

INTERVENTIONS:
Drug: Mercaptamine — Patients will be treated with 1 drop in each eye 4 times a day, at the same dose and regimen than the one indicated in adults and children from 2 years of age.

SUMMARY:
Cystadrops® is currently indicated in adults and children from 2 years of age diagnosed with cystinosis with corneal crystal accumulation observed.

However administration of Cystadrops® in patients below 2 years old could be of value for these patients and prevent the crystal deposit. It is the reason why as part of the Cystadrops® pediatric investigational plan (PIP), RECORDATI Rare Diseases committed to conduct a clinical study to assess Cystadrops® safety and efficacy in the pediatric population from 6 months to less than 2 years old.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged from 6 months to less than 2 years old
2. Cystinosis diagnosed patients confirmed by the physician and with presence of corneal cystine crystal deposits assessed during ophthalmic examination
3. Evidence of a signed and dated informed consent document indicating that parents/ legally acceptable representatives had been informed of all pertinent aspects of the study (if required by regulation)
4. Parents/ legally acceptable representatives who are willing to comply with regular visits and ophthalmic exams

Exclusion Criteria:

1. Contraindications to any of the Cystadrops® components
2. Participation in another ophthalmic investigational study or intent to participate during the course of the study
3. Any medical condition that would, in the opinion of the Investigator, interfere with the evaluation of the study objectives

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Ocular Serious Adverse Events, Serious Adverse Reactions related to Cystadrops, all Adverse Events that required discontinuation/withdrawal of IMP | Over a 90-day period
  To assess the safety profile of Cystadrops® over a 90-day period (ocular SAEs, SADRs)
Serious Adverse Reactions related to Cystadrops, all Adverse Events that required discontinuation/withdrawal of IMP | Over a 90-day period
  To assess the safety profile of Cystadrops® over a 90-day period (ocular SAEs, SADRs)
All Adverse Events that required discontinuation/withdrawal of IMP | Over a 90-day period
  To assess the safety profile of Cystadrops® over a 90-day period (ocular SAEs, SADRs)

SECONDARY OUTCOMES:
Ophtalmologic assessments (Best Corrected Visual Acuity) | 90-day period
  To assess the efficacy of Cystadrops® by measuring best corrected visual acuity (BCVA) of both eyes after 90 days of treatment with Cystadrops® when possible considering the age of the patients.
Ophtalmologic assessments (Corneal Cystine Crystal Score) | 90-day period
  To assess the efficacy of Cystadrops® by measuring Corneal cystine crystal score (CCCS), of both eyes after 90 days of treatment with Cystadrops® when possible considering the age of the patients.
Ophtalmologic assessments (Photophobia clinician-assessed evaluation according to a validated scale) | 90-day period
  To assess the efficacy of Cystadrops® by measuring photophobia of both eyes using a validated scale after 90 days of treatment with Cystadrops® when possible considering the age of the patients.

CONTACTS AND LOCATIONS:
Locations (6):
- UZ Leuven, Leuven, Belgium
- Hôpital Necker-Enfants Malades, Paris, France
- Klinik für Pädiatrische Nieren, Hanover, Germany
- Bambin Gesù Hospital in Palidoro, Roma, Italy
- United Kingdom (2):
  - Great Ormond Street Hospital, London
  - Manchester Royal Eye Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No